CLINICAL TRIAL: NCT02081729
Title: Assessment of VZV-specific ELISPOT Assay for Predicting VZV Infection in Kidney Transplant Recipients (AVE-KT)
Status: Terminated | Type: Observational
Why Stopped: low enrollment rate
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Advanced Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Assocaite Professor, Asan Medical Center
Other Study IDs: 2014-0107
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high VZV ELISPOT results: high spot counts in ELISPOT
- low VZV ELISPOT results: low spot counts in ELISPOT

SUMMARY:
VZV is one of the important opportunistic infection in transplant recipients.Until now, there is no laboratory method to stratify the risk of VZV reactivation after solid organ transplantation. Theoretically, VZV-specific cell-mediate immune response before solid organ transplantation will further categorize the patients into high or low risk of VZV development after solid organ transplantation. The investigators thus evaluate the usefulness of VZV-specific ELISPOT assay in kidney transplant candidates to predict the development of VZV infection after kidney transplantation.

DETAILED DESCRIPTION:
We will develop VZV-specific ELISPOT assay, then perform this assay before transplantation. We will evaluate whether this assay will predict zoster reactivation after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age 16 years or more
* agree with written informed consent
* WBC count 2000/uL or more

Exclusion Criteria:

* no exclusion criteria

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kindeny transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
zoster development | 6 months after transplantation

SECONDARY OUTCOMES:
mortality | 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea